CLINICAL TRIAL: NCT02862743
Title: Molecular Characterization of Advanced Stage Melanoma by Blood Sampling
Acronym: MELCIRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PO15097*
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

ARMS (1):
- patients with metastatic melanoma (Experimental): patients with metastatic melanoma (stage III unresectable or stage IV)
  Interventions: Other: patients with metastatic melanoma

INTERVENTIONS:
Other: patients with metastatic melanoma — Blood sample to realize molecular characterization of melanoma

SUMMARY:
Analysis of somatic mutations in tumors is currently indicated for daily practice in all metastatic melanoma. Actually, this research is limited to the mutation of three biomarkers validated by the l'Institut National du CAncer (INCA): BRAF, NRAS and CKIT. Moreover, in some cases it requires invasive biopsies.

In this context, molecular characterization of a tumor material flowing (circulating tumor DNA and / or circulating tumor cells) could afford to benefit patients in the best conditions of current targeted therapies and future.

DETAILED DESCRIPTION:
The main objective of this study will be to define the diagnostic sensitivity of a panel of biomarker on the circulating tumor DNA from peripheral blood.

The secondary objectives of this study will be:

* Study the concordance between mutations in circulating tumor DNA and mutations in tumor tissue - Study the associations between mutational profiles and clinical and histological features of melanoma.
* Study the prognostic impact on survival of the identified genetic profile from the circulating tumor DNA

ELIGIBILITY:
Inclusion Criteria:

* patient with melanoma confirmed histologically
* patient with metastatic melanoma (stage III unresectable or stage IV)
* patient consenting to participate to the study
* patient enrolled in the national healthcare insurance program
* patient older than 18 years

Exclusion Criteria:

- Metastatic tumor whose origin is doubtful (uncertain melanoma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of a panel of biomarker on the circulating tumor DNA from peripheral blood | Day 0
  Number of patients for which a circulating tumor DNA is detected (positivity of at least one marker of the panel)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Result] Beaudoux O, Riffaud L, Barbe C, Grange F. Prognostic factors and incidence of primary mucosal melanoma: a population-based study in France. Eur J Dermatol. 2018 Oct 1;28(5):654-660. doi: 10.1684/ejd.2018.3398. PMID 30378540